CLINICAL TRIAL: NCT06958393
Title: Effect of Opioid-free Anaesthesia on Postoperative Delirium in Elderly Patients Undergoing Gastrointestinal Surgery: a Single-centre, Prospective, Randomized Controlled Trial
Brief Title: Effect of Opioid-free Anaesthesia on Postoperative Delirium in Elderly Patients Undergoing Gastrointestinal Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Yongtao Sun, Professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: opioid-free anaesthesia
Record Dates: First submitted 2025-04-21; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Delirium - Postoperative; Opioid-Free Anaesthesia
Keywords: elderly patients; opioid-free anaesthesia; postoperative delirium; gastrointestinal surgery
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Esketamine; esmolol; Sufentanil; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-Based Anaesthesia (OBA) Group (Active Comparator): Patients receive conventional opioid-based general anaesthesia, including sufentanil and remifentanil during surgery and sufentanil-based patient-controlled intravenous analgesia (PCIA) postoperatively.
  Interventions: Drug: Sufentanil; Drug: Remifentanil
- Opioid-Free Anaesthesia (OFA) Group (Experimental): Patients receive opioid-free anaesthesia using a standardized multimodal regimen (dexmedetomidine, esmolol, and esketamine) for intraoperative management and esketamine-based PCIA postoperatively.
  Interventions: Drug: Dexmedetomidine; Drug: Esketamine; Drug: Esmolol

INTERVENTIONS:
Drug: Dexmedetomidine — Continuous infusion at 0.5-1.0 μg/kg/h during surgery
  Arms: Opioid-Free Anaesthesia (OFA) Group
Drug: Esketamine — Induction dose 0.3-0.5 mg/kg; maintenance 0.2-0.5 mg/kg/h; 0.02 mg/kg at closure; PCIA: 1.5 mg/kg in 100 mL saline
  Arms: Opioid-Free Anaesthesia (OFA) Group
Drug: Esmolol — Maintenance 20-100 μg/kg/min during surgery
  Arms: Opioid-Free Anaesthesia (OFA) Group
Drug: Sufentanil — 0.3-0.5 μg/kg induction; 0.15 μg/kg at closure; 2 μg/kg in 100 mL for PCIA
  Arms: Opioid-Based Anaesthesia (OBA) Group
Drug: Remifentanil — 0.2-1.0 μg/kg/min maintenance
  Arms: Opioid-Based Anaesthesia (OBA) Group

SUMMARY:
Background Postoperative delirium (POD) is a common acute and transient form of brain dysfunction in elderly patients following surgery that can lead to serious adverse clinical outcomes and even death. Although existing studies have preliminarily investigated the effects of opioid-free anaesthesia (OFA) on POD, high-quality evidence on these effects for elderly patients undergoing gastrointestinal surgery remains limited. This study aims to investigate the effects of OFA on the development of POD in elderly patients following gastrointestinal surgery.

Methods and analysis:

This single-centre, prospective, randomized controlled trial will be conducted at the First Affiliated Hospital of Shandong First Medical University, China. A total of 406 patients aged 65 years or older who are scheduled for elective gastrointestinal surgery will be randomly allocated to receive either opioid-free anaesthesia (OFA; dexmedetomidine, esmolol, and esketamine) or conventional opioid-based anaesthesia (OBA). The primary outcome is the incidence of POD 7 days after surgery. The secondary outcomes are all-cause mortality within 30 days after surgery, intraoperative haemodynamic changes, the 15-item quality of recovery (QoR-15) scores at 24 h, 48 h, and 72 h after surgery, complications during postoperative hospitalization, pain numerical rating scale (NRS) score at 72 h after surgery, incidence of nausea and vomiting at 72 h after surgery, morphine milligram equivalent for analgesics at 72 h after surgery, duration of anaesthesia (from induction to discontinuation), duration of surgery (from skin incision to the last suture), duration of post-anaesthesia care unit (PACU) stay, and length of hospital stay.

Discussion:

The results of this study may shed light on the effects of OFA on POD in elderly patients undergoing gastrointestinal surgery. The study is designed on the basis of the following key hypothesis: the use of opioid drugs for anaesthesia may increase the risk of POD through mechanisms such as blood-brain barrier destruction, neuroinflammatory responses, and central nervous system depression. Through the single-centre and prospective design of this randomized controlled trial, this study will directly analyse differences in the effects of OFA and conventional OBA on the incidence of POD, haemodynamic stability and long-term cognitive function in elderly patients.

gastrointestinal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years
2. American Society of Anesthesiologists (ASA) physical status classification I-III
3. Scheduled for elective gastrointestinal surgery under general anaesthesia
4. Body mass index (BMI) between 18.0 and 30.0 kg/m²

Exclusion Criteria:

1. Refusal to undergo surgery
2. Emergency surgery
3. Language impairment or severe hearing or visual deficits that hinder effective communication with research or surgical staff
4. History of neurological or psychiatric disorders, including Alzheimer's disease (AD), other forms of dementia, stroke, or psychosis
5. Long-term use of psychotropic medications (e.g., clozapine, risperidone, olanzapine, haloperidol, chlorpromazine)
6. Cardiac or craniocerebral surgery within the past year
7. Participation in other interventional clinical studies within the past 3 months
8. Preoperative cognitive impairment defined as a modified Telephone Interview for Cognitive Status (TICS-M) score ≤ 27
9. Patients will only be enrolled once, even if a subsequent surgery related to the primary procedure is performed

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-05-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of POD at discharge or within 7 days after surgery. | Discharge or within 7 days after surgery
  The proportion of participants who develop postoperative delirium, assessed either at discharge or within 7 days after surgery. Diagnosis of POD will be based on standardized clinical assessment tools (e.g., Confusion Assessment Method, CAM).Results will be reported as the percentage of participants (%).

SECONDARY OUTCOMES:
30-day All-Cause Mortality | Up to 30 days after surgery
  The proportion of participants who die from any cause during the initial hospitalization or within 30 calendar days following the index surgical procedure.The proportion of participants who die from any cause during the initial hospitalization or within 30 calendar days following the index surgical procedure. Results will be reported as the percentage of participants (%).

OTHER OUTCOMES:
Intraoperative Haemodynamic Changes | Intraoperative (from anesthesia induction to surgical closure)
  Changes in mean arterial pressure and heart rate recorded during surgery. Results will be reported as the mean change from baseline (mmHg or beats per minute).
Quality of Recovery-15 (QoR-15) Scores | 24, 48, and 72 hours after surgery
  QoR-15 scores assessed at 24 hours, 48 hours, and 72 hours after surgery. Results will be reported as the total score on the QoR-15 scale (range 0-150).
Postoperative Complications | From day of surgery through hospital discharge, up to 30 days
  Incidence of complications during postoperative hospitalization, including lung infection, urinary tract infection, cardiovascular and cerebrovascular accidents, abnormal liver function, postoperative bleeding, incision infection, deep venous thrombosis of the lower extremities, electrolyte imbalance, and hypoalbuminemia. Results will be reported as the percentage of participants (%).
Pain Numerical Rating Scale (NRS) Score at 72 Hours | 72 hours after surgery
  Pain intensity assessed using the NRS scale (0-10) at 72 hours after surgery. Results will be reported as the mean NRS score.
Incidence of Nausea and Vomiting at 72 Hours | 72 hours after surgery
  The proportion of participants experiencing nausea and/or vomiting at 72 hours after surgery. Results will be reported as the percentage of participants (%).
Morphine Milligram Equivalent (MME) Consumption for Analgesics at 72 Hours | 72 hours after surgery
  Total opioid consumption converted to morphine milligram equivalents (MME) at 72 hours after surgery. Results will be reported as total MME (mg).
Duration of Anaesthesia | From administration of anaesthetic agents to discontinuation of anaesthetic agents， up to 2 hours
  Time from induction of anaesthesia to discontinuation of anaesthetic agents. Results will be reported in minutes.
Duration of Surgery | From skin incision to completion of wound closure, up to 2 hours
  Time from skin incision to the last suture. Results will be reported in minutes.
Length of Stay in the Post-Anesthesia Care Unit (PACU) | From PACU admission to PACU discharge, measured in minutes, up to 60 minutes
  Time from arrival in the PACU to discharge from the PACU. Results will be reported in minutes.
Length of Hospital Stay | From day of surgery to hospital discharge, up to 30 days
  Total number of days from surgery to hospital discharge. Results will be reported in days.
Long-Term Cognitive Function at 6 Months | 6 months after surgery
  Cognitive function assessed at 6 months after surgery using standardized cognitive testing methods. Results will be reported as cognitive assessment scores.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

REFERENCES:
- [Derived] Du Y, Liu M, Yang X, Wu J, Gao X, Liu Q, Chen L, Sun X, Zhang M, Sun Y. Effect of opioid-free anaesthesia on postoperative delirium in elderly patients undergoing gastrointestinal surgery: study protocol for a single-centre, prospective, randomized controlled trial. BMC Geriatr. 2025 Jul 28;25(1):554. doi: 10.1186/s12877-025-06145-8. PMID 40721742